CLINICAL TRIAL: NCT00685087
Title: A Prospective Study of Natural History of Pancreatitis
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-Wiggins
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Chronic Pancreatitis
Keywords: To define the natural history and the clinical, laboratory and histomorphometric features of chronic pancreatitis (CP).; To identify clinical and laboratory parameters that correlate with the pathophysiologic state in patients with CP.; To quantify the behavioral abnormalities associated with CP.; To determine psychological and behavioral correlates of CP disease progression and outcomes.
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To prospectively define the natural history and the clinical, laboratory and histomorphometric features of chronic pancreatitis (CP) of varying etiology. To identify clinical and laboratory parameters that correlate with the pathophysiologic state in patients with CP. To quantify the behavioral abnormalities associated with CP. To determine psychological and behavioral correlates of CP disease progression and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with pancreatitis

Exclusion Criteria:

* Lack of consent, age <18 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects presenting to the Pancreatitis clinic with diagnosis of pancreatitis
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2004-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bimaljit S Sandhu, M.D, Principal Investigator — Virginia Commonwealth University Medical Center, Richmond VA 23298
Locations (1):
- Virginia Commonwealth University Medical center, Richmond, Virginia, United States

REFERENCES:
- [Derived] Sandhu B, Vitazka P, Ferreira-Gonzalez A, Pandya A, Vachhani R, Bouhaidar D, Zfass A, Sanyal A. Presence of SPINK-1 variant alters the course of chronic pancreatitis. J Gastroenterol Hepatol. 2011 Jun;26(6):965-9. doi: 10.1111/j.1440-1746.2011.06713.x. PMID 21375584